CLINICAL TRIAL: NCT00953303
Title: The Effects of Glucocorticoids on Mortality and Renal Function in Patients With Acute Decompensated Heart Failure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Kun-shen Liu M.D., Professor, Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hebmu 08-12B
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Heart Failure
Keywords: heart failure; prednisone; cardiovascular mortality; renal function
MeSH Terms: conditions — Heart Failure | interventions — Glucocorticoids; dexamethasone 21-phosphate; Prednisone; Standard of Care; Furosemide; Torsemide; Nitroglycerin; Dopamine; Dobutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- glucocorticoid (Experimental)
  Interventions: Drug: glucocorticoid
- Standard care (Active Comparator)
  Interventions: Drug: standard care

INTERVENTIONS:
Drug: glucocorticoid — One dose of Dexamethasone (20mg/day) followed by prednisone 1mg/kg/day with a maximum dose of 60mg/day.
  Other Names: Dexamethasone Sodium Phosphate; prednisone acetate tablets
  Arms: glucocorticoid
Drug: standard care — The patients will be given standard care such as diuretics, inotropic and/or vasodilator in acute decompensated congestive heart failure management.
  Other Names: Furosemide; torsemide; nitroglycerin; dopamine; Dobutamine
  Arms: Standard care

SUMMARY:
Evidence showed that glucocorticoids could induce potent diuretic actions and improve renal functions in patients with decompensated congestive heart failure. Thus we design this study to determine the efficacy of glucocorticoids on cardiovascular mortality in the 30 days following randomization.

DETAILED DESCRIPTION:
Newly emerging clinical evidence showed glucocorticoids, when added to best conventional therapy, could produce potent diuretic effects, and improve renal functions in patients with decompensated congestive heart failure. It holds ture even in the patients who failed to respond to high dose of furosemide (>200mg/day). The present study is to confirm the clinical efficacy of glucocorticoids on cardiovascular mortality in patients with decompensated congestive heart failure who are on best conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dyspnea at rest due to acutely decompensated CHF requiring hospitalization and intravenous therapy. The cardiac etiology for acutely decompensated CHF was established by echocardiogram and/or a chest x-ray film and 2 of the following:

  1. >2-pillow orthopnea before study entry
  2. Jugular venous distention and/or abdominal discomfort due to mesenteric congestion.

Patients may have had acute decompensation of chronic heart failure, gradual worsening of chronic heart failure, or new onset of acutely decompensated CHF. Patients who were receiving intravenous therapy i.e. Inotropic and/or vasodilator but who otherwise met entry criteria were also permitted into the study. Patients with signs of cardiac shock were also permitted into the study.

Exclusion Criteria:

* Patient refusal
* Any signs of infection
* any condition that would contraindicate a glucocorticoids use
* Poor controlled hypertension
* Poor controlled diabetes mellitus
* Active myocarditis
* Malignancy or other terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-01; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular mortality in the 30 days following randomization. | 30 days following randomization

SECONDARY OUTCOMES:
Renal function | on day 7
physician assessed global clinical status | on day 3 and day 7
patient assessed dyspnea | on day 3 and day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Kunshen Liu, MD, Principal Investigator — The First Hospital of Hebei Medical University
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China